CLINICAL TRIAL: NCT02174367
Title: An Observational Cohort Study to Evaluate Factors Affecting Prevalence of Fatty Liver Disease and Fibrosis and Factors Affecting Response to Treatment in Patients With Psoriasis
Brief Title: An Observational Cohort Study Evaluating Fatty Liver Disease and Liver Fibrosis in Moderate to Severe Psoriasis
Acronym: CORE
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: King's College London (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: WS1851782; 11/LO/1236 (Other: London REC reference number)
Record Dates: First submitted 2014-05-22; First posted 2014-06-25 (Estimated); Last update posted 2017-08-04 (Actual); Status verified 2017-06

CONDITIONS: Psoriasis Chronic; Liver Fibrosis; Fatty Liver; Non-alcoholic Fatty Liver Disease
Keywords: Chronic plaque psoriasis; Liver fibrosis; Fatty liver disease; Non-alcoholic fatty liver disease; Transient elastography; Fibroscan; Procollagen-3 N-Terminal peptide; Alanine aminotransferase; Liver function tests
MeSH Terms: conditions — Liver Cirrhosis; Fatty Liver; Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum stored for analysis of non-invasive markers of fibrosis and DNA analysis
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Psoriasis: Patients with moderate to sever psoriasis attending a tertiary referral center. patients will be evaluated with a questionnaire, measurement of height,weight, waist circumference, fasting bloods, abdominal ultrasound and transient elastography.
  Interventions: Device: Transient elastography

INTERVENTIONS:
Device: Transient elastography — a noninvasive tool for measuring liver stiffness as a predictor of liver fibrosis
  Other Names: Fibroscan

SUMMARY:
• Main objectives and outcome measures.

1. Establish prevalence of and factors contributing to fatty liver disease and liver fibrosis in patients with psoriasis.

   Fatty liver disease diagnosed via ultrasound. Liver fibrosis diagnosed by liver biopsy or non-invasive tests of fibrosis including transient elastography, ultrasound, serum markers of fibrosis including procollagen-3-N-terminal peptide (P3NP).
2. Evaluate non-invasive markers of liver fibrosis in the psoriasis population. Namely transient elastography, standard liver function tests and P3NP.
3. Evaluate the impact of psoriasis disease severity and comorbidities including metabolic syndrome on response to treatment in patients with psoriasis.

Data on co-morbid disease collected through questionnaires and review of medical records. Response to treatment assessed using psoriasis area and severity index (PASI) physician global assessment (PGA) and dermatology life quality index (DLQI).

* Study population: 380 patients with moderate to severe psoriasis will be prospectively recruited to the study.
* Chief investigator: Professor Jonathan Barker. Co-investigator: Professor Catherine Smith
* Sponsor/funding organization: Pfizer and Biomedical Research Centre (BRC) at Guys and St Thomas Hospitals Trust

ELIGIBILITY:
Inclusion Criteria:

* Patients who have given written informed consent
* Psoriasis patients - chronic plaque-type psoriasis; PASI of 10 or above currently or in past.
* 18 yrs. of age

Exclusion Criteria:

* Patients who have not given written informed consent
* Patients under 18 yrs. of age
* Patients with a PASI less than 10.
* Pregnant women

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospital outpatient clinic
Sampling Method: Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2012-11 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
Number of participants with liver fibrosis. | 12 months after enrollment
  Liver fibrosis will be assessed by transient elastography and the use of standard liver function tests and other serum markers of fibrosis including P3NP. In a minority of cases fibrosis will be diagnosed by liver biopsy and evaluation of histology. Risk factors for the development of fibrosis including metabolic syndrome, alcohol and methotrexate use will be evaluated.

SECONDARY OUTCOMES:
Number of participants with fatty liver disease diagnosed by ultrasound | Within 12 months of enrollment
  Fatty liver disease will be defined by the presence or absence of fatty changes on abdominal ultrasound. Risk factors for the development of fatty liver disease including abdominal obesity, diabetes, and alcohol use will be evaluated.

OTHER OUTCOMES:
Sensitivity, specificity, and likelihood ratios of noninvasive tests of liver fibrosis | Within 12 months of enrollment
  The performance of non-invasive markers of fibrosis including standard liver function tests, P3NP, transient elastography and abdominal ultrasound will be assessed in this cohort of patients with chronic plaque psoriasis.
Response to treatment measured by PASI and PGA scores | 12-24 months following enrollment
  Response to treatment will be measure by physician global assessment (PGA) PASI and DLQI. Factors assessed include demographic data, psoriasis disease history, co-morbid disease and family history assessed by questionnaire. Lipid and glycaemic status assessed by fasting bloods.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan N Barker, BSC MD FRCP, Principal Investigator — King's College London; Catherine H Smith, MD FRCP, Study Director — Guys and St Thomas' Hospitals Foundation Trust and King's College London
Locations (1):
- Guys and St Thomas NHS Foundation trust and King's College London, London, United Kingdom

REFERENCES:
- [Background] Maybury CM, Jabbar-Lopez ZK, Wong T, Dhillon AP, Barker JN, Smith CH. Methotrexate and liver fibrosis in people with psoriasis: a systematic review of observational studies. Br J Dermatol. 2014 Jul;171(1):17-29. doi: 10.1111/bjd.12941. Epub 2014 Jul 15. PMID 24606161
- [Background] Maybury CM, Samarasekera E, Douiri A, Barker JN, Smith CH. Diagnostic accuracy of noninvasive markers of liver fibrosis in patients with psoriasis taking methotrexate: a systematic review and meta-analysis. Br J Dermatol. 2014 Jun;170(6):1237-47. doi: 10.1111/bjd.12905. PMID 24588075
- [Background] Samarasekera EJ, Smith CH; National Institute of Health and Care Excellence; Royal College of Physicians. Psoriasis: guidance on assessment and referral. Clin Med (Lond). 2014 Apr;14(2):178-82. doi: 10.7861/clinmedicine.14-2-178. PMID 24715130
- [Background] Smith CH, Barker JN. Psoriasis and its management. BMJ. 2006 Aug 19;333(7564):380-4. doi: 10.1136/bmj.333.7564.380. No abstract available. PMID 16916825
- [Background] Nestle FO, Kaplan DH, Barker J. Psoriasis. N Engl J Med. 2009 Jul 30;361(5):496-509. doi: 10.1056/NEJMra0804595. No abstract available. PMID 19641206
- [Background] Boehncke WH, Boehncke S, Schon MP. Managing comorbid disease in patients with psoriasis. BMJ. 2010 Jan 15;340:b5666. doi: 10.1136/bmj.b5666. No abstract available. PMID 20080817
- [Background] Fonia A, Jackson K, Lereun C, Grant DM, Barker JN, Smith CH. A retrospective cohort study of the impact of biologic therapy initiation on medical resource use and costs in patients with moderate to severe psoriasis. Br J Dermatol. 2010 Oct;163(4):807-16. doi: 10.1111/j.1365-2133.2010.09944.x. PMID 20662837
- [Derived] Maybury CM, Porter HF, Kloczko E, Duckworth M, Cotton A, Thornberry K, Dew T, Crook M, Natas S, Miquel R, Lewis CM, Wong T, Smith CH, Barker JN. Prevalence of Advanced Liver Fibrosis in Patients With Severe Psoriasis. JAMA Dermatol. 2019 Sep 1;155(9):1028-1032. doi: 10.1001/jamadermatol.2019.0721. PMID 31166567